CLINICAL TRIAL: NCT06772714
Title: Long Term Follow-up of the Ponto Wide Implant: 10 Years of Clinical Evaluation
Brief Title: 10-year Follow-up of the Ponto Wide-implant
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Center Nijmegen (Other)
Collaborators: Oticon Medical (Industry)
Responsible Party: Principal Investigator, Carine Hajema, Investigator, University Medical Center Nijmegen
Other Study IDs: 2024-17533
Record Dates: First submitted 2024-12-20; First posted 2025-01-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Survival of the Ponto Wide Implant
Keywords: Implant survival; Ponto Wide implant; Oticon; 10 years; Deafness; Hearing loss; Hearing disorders
MeSH Terms: conditions — Deafness; Hearing Loss; Hearing Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a Ponto Wide Implant for 10 years: The study population consists of patients who received a Ponto Wide implant (4.5 mm diameter, 4.0 mm length) at least 10 years ago. Only patients who participated in one of the two previous completed studies (Long-term stability and survival rates of a novel Oticon Medical bone conduction device implant, Three-year Outcomes of a Randomized Controlled Trial Comparing a 4.5-mm-Wide to a 3.75-mm-Wide Titanium Implant for Bone Conduction Hearing) will be included

SUMMARY:
The goal of this single center, prospective study is to investigate the survival of the Ponto Wide Implant at least 10 years after implantation.

Secondary objectives are:

1. To determine the amount and causes of implant loss and implant and/or abutment removal.
2. To establish the stability of the implant.
3. To assess skin complications.
4. To investigate daily usage and the number of hours of use of the sound processor.
5. To determine the quality of life.

During a check-up of the implant at the outpatient clinic, the skin around the implant will be assessed, the stability of the implant will be measured, and the patient will be asked to complete two questionnaires.

DETAILED DESCRIPTION:
Patients who participated in the previous studies concerning the Ponto Wide implant from Oticon (3 years after implantation) will be approached. If consent is given, they will be added to the database of the already completed studies, and new data will be stored in the same database. The patients were already pseudonymized in the previous studies, and the database is secured with a code that is only accessible to individuals directly involved in the research

ELIGIBILITY:
Inclusion Criteria:

* Implantation with Ponto Wide implant (diameter 4.5 mm, length 4.0 mm)
* Ten or more years of post-operative follow-up.
* Valid informed consent

Exclusion Criteria:

* No specific exclusion criteria have been set for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients who received a Ponto Wide implant (4.5 mm diameter, 4.0 mm length) at least 10 years ago and previously participated in one of two already completed studies.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Implant survival | It will be assessed during the clinic visit between November 2024 and March 2025.
  The number of Ponto Wide implants that have survived 10 years after implantation.

SECONDARY OUTCOMES:
Amount of implant loss | This will be examined during the period from November 2024 to March 2025
  The number of implant losses over the past 10 years based on the patient files.
Reasons of implant loss | This will be examined during the period from November 2024 to March 2025
  The reason for each implant loss.
Amount of abutment loss | This will be examined during the period from November 2024 to March 2025
  The number of abutment losses over the past 10 years based on the patient files.
Reasons of abutment loss | This will be examined during the period from November 2024 to March 2025
  The reason for each abutment loss.
Amount of implant removal | This will be examined during the period from November 2024 to March 2025
  The number of implant removal over the past 10 years based on the patient files.
Reasons of implant removal | This will be examined during the period from November 2024 to March 2025
  The reason for each implant removal.
Amount of abutment removal | This will be examined during the period from November 2024 to March 2025
  The number of abutment removals over the past 10 years based on the patient files.
Reasons of abutment removal | This will be examined during the period from November 2024 to March 2025
  The reason for each abutment removal.
Implant stability Quotient (ISQ) measured using Osstell | It will be assessed during the clinic visit between November 2024 and March 2025.
  ISQ (implant Stability Quotient) is a measurement scale for use with the Resonance Frequency Analysis (RFA) method of determining implant stability. The measurement is made using the Osstell Mentor equipment (Osstell, Sweden) with SmartPegs. ISQ values range from 1 to 100, the higher the score the higher the stability. The highest and lowest score obtained from perpendicular measurements will be registered.
Skin complication | It will be assessed during the clinic visit between November 2024 and March 2025.
  Skin complication rates at >10-year follow-up are assessed using both the Holgers classification and the IPS-score. Both classification systems are standardized scales to clinically assess the skin condition around the implant.
Sound processor use | It will be assessed during the clinic visit between November 2024 and March 2025.
  Average sound processor usage (hours per day; days/week) >10 years post-surgery.
Glasgow Benefit Inventory (GBI) | It will be assessed during the clinic visit between November 2024 and March 2025.
  The GBI questionnaire is used to evaluate the quality of life after a medical intervention. The questionnaire consists of 18 items corresponding to different aspects of the patient's well-being: quality of life, self-confidence, support, general health, and social involvement. The scoring ranges from 1 to 5, indicating that a higher score means the statement is more applicable to the patient after the intervention.
International Outcome Inventory for Hearing Aids (IOI-HA) | It will be assessed during the clinic visit between November 2024 and March 2025.
  The IOI-HA questionnaire is a seven-item tool designed to be broadly applicable in evaluating the effectiveness of hearing aid treatments. These questions provide insight into how satisfied patients are with their hearing aids. Each statement offers five possible responses on an ascending scale, indicating whether the answer is more or less applicable to the statement.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Myalnus, Prof. dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kruyt IJ, Kok H, Bosman A, Nelissen RC, Mylanus EAM, Hol MKS. Three-Year Clinical and Audiological Outcomes of Percutaneous Implants for Bone Conduction Devices: Comparison Between Tissue Preservation Technique and Tissue Reduction Technique. Otol Neurotol. 2019 Mar;40(3):335-343. doi: 10.1097/MAO.0000000000002105. PMID 30742596
- [Background] den Besten CA, Bosman AJ, Nelissen RC, Mylanus EA, Hol MK. Controlled Clinical Trial on Bone-anchored Hearing Implants and a Surgical Technique With Soft-tissue Preservation. Otol Neurotol. 2016 Jun;37(5):504-12. doi: 10.1097/MAO.0000000000000994. PMID 26945315
- [Background] Nelissen RC, den Besten CA, Mylanus EA, Hol MK. Stability, survival, and tolerability of a 4.5-mm-wide bone-anchored hearing implant: 6-month data from a randomized controlled clinical trial. Eur Arch Otorhinolaryngol. 2016 Jan;273(1):105-11. doi: 10.1007/s00405-015-3593-x. Epub 2015 Mar 20. PMID 25790770
- [Background] Vijverberg MA, Caspers CJI, Kruyt IJ, Mylanus EAM, Hol MKS. Prospective 5 year outcomes of different implant designs and surgical techniques in 68 patients with bone anchored hearing implants. Clin Otolaryngol. 2023 Jan;48(1):65-69. doi: 10.1111/coa.13974. Epub 2022 Sep 17. No abstract available. PMID 36054740
- [Background] Kruyt IJ, Nelissen RC, Mylanus EAM, Hol MKS. Three-year Outcomes of a Randomized Controlled Trial Comparing a 4.5-mm-Wide to a 3.75-mm-Wide Titanium Implant for Bone Conduction Hearing. Otol Neurotol. 2018 Jun;39(5):609-615. doi: 10.1097/MAO.0000000000001761. PMID 29561377

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT06772714/Prot_SAP_000.pdf